CLINICAL TRIAL: NCT03692624
Title: Use of Heart Rate Variability (HRV) Biofeedback for Symptom Management Among Cancer Survivors: Pilot Intervention
Brief Title: Use of Heart Rate Variability (HRV) Biofeedback for Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Collaborators: University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00042898
Record Dates: First submitted 2018-09-27; First posted 2018-10-02 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Cancer
Keywords: cancer survivors; heart rate variability; biofeedback
MeSH Terms: conditions — Neoplasms | interventions — Biofeedback, Psychology

STUDY DESIGN:
Intervention Model Description: Cancer patients will be recruited from the Cancer Institute at Greenville Health System. Random assignment to the HRV-B or control group will occur after baseline assessment. During the baseline assessment, participants will be asked to fill out a questionnaire, including information about symptoms and feelings. Participant heart rate (pulse) and breathing will be measured for 15 minutes. Baseline heart rate will be measured with a sensor loosely attached to the wrist. Breathing will be monitored by another sensor attached around the abdomen by a belt. Each weekly HRV-B training session will last 30-45 minutes. In each session, heart rate and breathing will be monitored while the participant is viewing pleasant images on a computer screen. An Intervention professional will be present throughout the session. While viewing the images, the participant will be coached on how to control their pulse.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Biofeedback. Participants receiving the HRV-B intervention will complete a baseline assessment, a minimum of 4 weeks and up to 6 weekly training sessions (until the criterion of HRV coherence is met), and a final appointment (3-7 days later) where post-training HRV and symptom inventories will be recorded.
  Interventions: Behavioral: Biofeedback
- Control Group (No Intervention): To control for the laboratory environment or other potential placebo effects, a control group will receive their usual follow-up care for their cancer diagnosis and will complete baseline and post-baseline outcome assessments without any HRV-B training.

INTERVENTIONS:
Behavioral: Biofeedback — Heart Rate Variability Biofeedback
  Arms: Intervention Group

SUMMARY:
Heart rate variability biofeedback (HRV-B) is a complementary, non-pharmacologic therapy that is being tested to see if it can help cancer survivors reduce their symptoms of pain, stress, insomnia, fatigue, or depression. HRV-B is an interactive procedure in which participants relax and breathe regularly while watching the a computer screen. The computer screen provides feedback that helps people increase their heart rate variability.

DETAILED DESCRIPTION:
Cancer survivors often suffer from prolonged and persistent symptom clusters that can include: pain, stress, depression, fatigue, and insomnia; symptoms that have each been associated with inflammation. The number of cancer survivors in the United States is expected to triple by the year 2030. Thus, there is a compelling need to develop and refine effective methods to promote high quality cancer survivorship. Dysregulation of autonomic function is a key pathophysiological 'common denominator' whereby many cancer-related symptoms likely converge. Heart rate variability (HRV) is a valid, noninvasive measure of autonomic function with established pathological and psychophysiological attributes. Reduced HRV is a known mortality risk factor, and about 80% of advanced cancer patients exhibit autonomic dysregulation. Cancer survivors with reduced HRV have increased mortality risk relative to those with normal HRV. HRV biofeedback (HRV-B) is an interactive procedure whereby patients learn to increase HRV and restore autonomic balance. HRV coherence refers to a state of optimum HRV rhythm that produces physiological entrainment of HRV, respiration, and the baroreflex. With HRV coherence, consecutive inter-beat intervals cycle from maximum to minimum and back to maximum over a period of about 10 seconds, which is associated with increased parasympathetic and decreased sympathetic tone, and a heightened state of well-being including improved affect, cognition, and executive function. Previous research suggests that HRV-B interventions may be useful for reducing symptoms of: chronic pain, anxiety, depression, post-traumatic stress disorder (PTSD), heart disease, and insomnia. HRV-B thus represents a promising complementary, nonpharmacological therapy that merits examination for relief of chronic pain and related symptoms among cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* histopathologically confirmed diagnosis of cancer having completed radiation or chemotherapy
* 18 years of age or older
* English literate

Exclusion Criteria:

* patients receiving concurrent treatment for cancer except hormonal or biologic therapy
* patients with cardiovascular disorders that affect HRV parameters (paroxysmal supraventricular tachycardia, atrial fibrillation, myocardial infarction within 12 months, unstable angina)
* patients receiving medications that affect cardiac rhythm (angiotensin converting enzyme, calcium channel, or beta-adrenergic inhibitors)
* patients with a pacemaker or defibrillator
* patients who have had a heart transplant or by-pass surgery within 1 year
* patients with any active seizure disorder or use of antiseizure or anticonvulsant medication prescribed specifically for seizure disorder
* patients with a pre-existing dementia prior to cancer diagnosis
* patients with a moderate (without good recovery) or severe head injury or stroke in last 6 months
* patients with evidence of active substance abuse or dependence
* patients with a history of any major psychiatric disorder
* patients with a history of brain metastases, primary brain cancer, or altered cognitive abilities
* patients with any use of long acting (extended release) opioid medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-05-10 (Actual); Primary Completion 2017-04-19 (Actual); Study Completion 2020-02-07 (Actual)

PRIMARY OUTCOMES:
Reduced Pain | Weekly for 4 to 6 weeks
  Participants will attend an HRV-B training session once a week for up to 6 weeks. They will complete a questionnaire which includes a symptom cluster assessment related to pain using the Brief Pain Inventory (BPI).
Reduced Stress | Weekly for 4 to 6 weeks
  Participants will attend an HRV-B training session once a week for up to 6 weeks. They will complete a SUSCRO Distress Inventory which includes a symptom cluster inventory related to distress. The inventory includes 12 questions which are self-rated from 0 (not at all) to 4 (most of the time). Lower scores indicate less distress and higher scores indicate severe distress.
Reduced Fatigue | Weekly for 4 to 6 weeks
  Participants will attend an HRV-B training session once a week for up to 6 weeks. They will complete a questionnaire which includes a symptom cluster inventory related to fatigue using the Multi-Dimensional Fatigue Inventory (MFI).
Reduced Depression | Weekly for 4 to 6 weeks
  Participants will attend an HRV-B training session once a week for up to 6 weeks. They will complete a questionnaire which includes a symptom cluster inventory related to depression using the Beck Depression Inventory II (BDI-II).
Reduced Insomnia | Weekly for 4 to 6 weeks.
  Participants will attend an HRV-B training session once a week for up to 6 weeks. They will complete the Insomnia Symptom Questionnaire (ISQ) which includes a symptom cluster inventory related to sleep patterns. The inventory includes 13 self-rated questions. Questions 1, 2 or 5 are used to determine the presence, frequency and duration of sleep symptom criteria. Questions 6 through 13 are used to identify significant daytime consequences of sleep disturbance.

CONTACTS AND LOCATIONS:
Overall Officials: Mark A O'Rourke, MD, Principal Investigator — Prisma Health-Upstate
Locations (1):
- Greenville Health System Cancer Institute, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Information published will only be done in aggregate. All participant information will be de-identified.

REFERENCES:
- [Background] Kim DH, Kim JA, Choi YS, Kim SH, Lee JY, Kim YE. Heart rate variability and length of survival in hospice cancer patients. J Korean Med Sci. 2010 Aug;25(8):1140-5. doi: 10.3346/jkms.2010.25.8.1140. Epub 2010 Jul 21. PMID 20676323
- [Background] Hoffmann J, Grimm W, Menz V, Wied M, Sprenger A, Arnold R, Maisch B. Prognostic value of heart rate variability analysis in patients with carcinoid syndrome. Digestion. 2001;63(1):35-42. doi: 10.1159/000051870. PMID 11173898
- [Background] de Miguel Sanchez C, Elustondo SG, Estirado A, Sanchez FV, de la Rasilla Cooper CG, Romero AL, Otero A, Olmos LG. Palliative performance status, heart rate and respiratory rate as predictive factors of survival time in terminally ill cancer patients. J Pain Symptom Manage. 2006 Jun;31(6):485-92. doi: 10.1016/j.jpainsymman.2005.10.007. PMID 16793488
- [Background] Mouton C, Ronson A, Razavi D, Delhaye F, Kupper N, Paesmans M, Moreau M, Nogaret JM, Hendlisz A, Gidron Y. The relationship between heart rate variability and time-course of carcinoembryonic antigen in colorectal cancer. Auton Neurosci. 2012 Jan 26;166(1-2):96-9. doi: 10.1016/j.autneu.2011.10.002. Epub 2011 Nov 9. PMID 22070982
- [Background] Appelhans BM, Luecken LJ. Heart rate variability and pain: associations of two interrelated homeostatic processes. Biol Psychol. 2008 Feb;77(2):174-82. doi: 10.1016/j.biopsycho.2007.10.004. Epub 2007 Oct 12. PMID 18023960
- [Background] Kapitza KP, Passie T, Bernateck M, Karst M. First non-contingent respiratory biofeedback placebo versus contingent biofeedback in patients with chronic low back pain: a randomized, controlled, double-blind trial. Appl Psychophysiol Biofeedback. 2010 Sep;35(3):207-17. doi: 10.1007/s10484-010-9130-1. PMID 20237953
- [Background] Berry ME, Chapple IT, Ginsberg JP, Gleichauf KJ, Meyer JA, Nagpal ML. Non-pharmacological Intervention for Chronic Pain in Veterans: A Pilot Study of Heart Rate Variability Biofeedback. Glob Adv Health Med. 2014 Mar;3(2):28-33. doi: 10.7453/gahmj.2013.075. PMID 24808979
- [Derived] Burch JB, Ginsberg JP, McLain AC, Franco R, Stokes S, Susko K, Hendry W, Crowley E, Christ A, Hanna J, Anderson A, Hebert JR, O'Rourke MA. Symptom Management Among Cancer Survivors: Randomized Pilot Intervention Trial of Heart Rate Variability Biofeedback. Appl Psychophysiol Biofeedback. 2020 Jun;45(2):99-108. doi: 10.1007/s10484-020-09462-3. PMID 32358782